CLINICAL TRIAL: NCT04172766
Title: Apple Hearing Study: Characterization of Headphone Audio Levels, and Optional Wristwatch-Based Environmental Sound Levels, with Variable User Interface
Brief Title: Apple Hearing Study
Acronym: AHS
Status: Recruiting | Type: Observational
Sponsor: Apple Inc. (Industry)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Richard Neitzel, Associate Professor of Environmental Health Sciences and Associate Professor of Global Public Health, University of Michigan
Other Study IDs: Pro00037864; HUM00167885 (Other: University of Michigan IRB)
Record Dates: First submitted 2019-11-13; First posted 2019-11-21 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Hearing Loss, Noise-Induced; Hearing Loss; Tinnitus
Keywords: Hearing Loss; Noise Exposure; Noise Induced Hearing Loss; Listening Volume; Environmental Noise; Music; Audiometry; Speech-in-Noise; Hearing Ability; Headphones; Headphone audio level; Ambient noise; Occupational noise; Heart rate; Tinnitus
MeSH Terms: conditions — Hearing Loss, Noise-Induced; Hearing Loss; Tinnitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort: Participants will be asked to read and sign the study ICF within the app if they agree and are willing to participate. After providing informed consent to participate, participants will be directed to select which data they want to share from the Health App via HealthKit and SensorKit to the Research app. All Research app users are asked to complete contact information and demographic questions that may be common across multiple Research app studies, such as age, race, sex, location of residence, and socioeconomic status. Participants will be asked to complete surveys approximately every other month for a total of about 1.5 hours over the entire year. Participants will be asked to complete three types of hearing tests 2-6 times per year; Interactive Tinnitus Tasks, Pure Tone Audiometry, and Speech in Noise. Participants will also be requested to complete brief on-demand surveys following high sound level measurements from headphones or the watch, at most monthly.

SUMMARY:
The Apple Hearing Study is a partnership between the University of Michigan and Apple to study sound exposure and its impact on hearing health. This groundbreaking study will advance the understanding of how hearing could be impacted over time by exposure to sound at certain levels. The investigators will measure headphone and environmental sound exposures over time among participants, and determine how these exposures impact hearing and stress levels. US residents who own an iPhone, download the Apple Research app and consent to participate will be randomly assigned to two groups, one with a "Basic" user interface in the Research app, and one with an "Advanced" user interface. Users in the "Advanced" group will receive additional information about their exposures and be given additional surveys and hearing tests based on their music and environmental sound exposures. The study will provide investigators with a better understanding of listening behavior and its overall impact on hearing health. This information will in turn help guide public health policy and prevention programs designed to protect and promote hearing health in the US and globally.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of eligibility screening, ascertained from self-reported date of birth. Potential subjects in the states of Alabama and Nebraska must be 19 or older (legal age of consent in these states), and 21 and older for any subjects in Puerto Rico.
* Live in the United States of America at time of eligibility screening, ascertained from self-report.
* Proficient in written and spoken English, defined by self-report.
* Participants must NOT share their iCloud account, iPhone or other devices such as Apple Watch with anyone else as this would make it challenging for researchers to use their information.
* Possession of the following, ascertained from automatic hardware/software/device pairing check:

  * iPhone with iOS versions capable of supporting the Research app used to complete screening eligibility.
  * Optional: Apple Watch (any model) paired with iPhone; an Apple Watch Series 4 or later is required to share environmental sound levels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults age 18 or older that live in the U.S. or U.S. territories and have iPhone with the Research app installed.
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Headphone audio level patterns | From enrollment to the end of followup at 10 years
  For the entire cohort over various timeframes
Difference in Headphone Audio Level patterns | From enrollment to the end of followup at 10 years
  This will include assessment of sound pressure level and time at baseline and over the duration of the study.
Association between Headphone Audio Level patterns and Pure Tone Audiometry | From enrollment to the end of followup at 10 years
  Analysis will occur for each tested frequency (dB HL at 125 Hz, 250 Hz, 500 Hz, 1 kHz, 2 kHz, 4kHz, and 8 kHz assessed for both ears) for both ears at baseline and over the duration of the study.
Association between Headphone Audio Level patterns and Speech in Noise | From enrollment to the end of followup at 10 years
  Analysis will assess the speech recognition threshold and it's relationships with HAL at baseline and over the duration of the study
Association between Headphone Audio Level patterns and tinnitus matching | From enrollment to the end of followup at 10 years
  At baseline and over the duration of the study
Association between general health and individual characteristics and sound levels and/or audiometry tasks | From enrollment to the end of followup after 10 years
  Headphone Audio Levels will be assessed as the sound level and the audiometry tasks assessed will be Pure Tone Audiometry, Speech in Noise, and tinnitus matching
Change from baseline to final audiometry | From enrollment to the end of followup after 10 years
  Including both Pure Tone Audiometry and Speech in Noise
Change from baseline in abbreviated Pure Tone Audiometry following high headphone audio level notification | From enrollment to the end of followup after 10 years
  This comparison will occur for two frequencies (1 kHz and 4 kHz for both ears) within 24 hours of acute loud Headphone Audio Level exposure (LEQ equivalent to >97 dBA for >30 minutes)
Headphone Audio Level association with baseline survey questions | From enrollment to the end of followup after 10 years
  This will includes questions about typical headphone us, typical environmental exposures, and hearing ability.
Baseline Audiometry association with baseline survey questions | From enrollment to the end of followup after 10 years
  Baseline Audiometry includes both Pure Tone Audiometry and Speech in Noise. Survey questions include those regarding typical headphone use, typical environmental exposures, and hearing ability.
Final Audiometry association with end-of-study survey questions | At the end of followup after 10 years
  Final Audiometry includes Pure Tone Audiometry and Speech in Noise. The end-of-study survey questions include typical headphone use, typical environmental exposures, and hearing ability.
Change in survey questions | From enrollment to the end of followup after 10 years
  Survey questions regarding exposure changes over the course of the study
Association between hearing ability and changes in hearing health and related health conditions | From enrollment to the end of followup after 10 years
  Hearing ability is evaluated both as perceived and evaluated. Changes in hearing health include audiometry and tinnitus. Related health conditions include items such as cognition, sleep, mental health, activity, mobility, and more.
Descriptive assessment of participant use and experience | From enrollment to the end of followup after 10 years
  Experience with hearing related tools and device

SECONDARY OUTCOMES:
Difference in Environmental Sound Level Patterns | From enrollment to the end of followup after 10 years
  Including sound pressure level and time at baseline and over the duration of the study. This outcome is only among participants that use Apple Watch.
Association between Headphone Audio Levels and Environmental Sound Level patterns | From enrollment to the end of followup after 10 years
  This outcome is only among participants that use Apple Watch.
Association between Environmental Sound Level patterns and Pure Tone Audiometry. | From enrollment to the end of followup after 10 years
  At baseline and over the duration of the study. This outcome is only among Participants that use Apple Watch.
Association between Environmental Sound Level patterns and Speech in Noise | From enrollment to the end of followup after 10 years
  At baseline and over the duration of the study. This outcome is only among Participants that use Apple Watch.
Association between Environmental Sound Level patterns and tinnitus matching task | From enrollment to the end of followup after 10 years
  At baseline and over the duration of the study. This outcome is only among Participants that use Apple Watch.
Association between general health and personal characteristics and sound levels and hearing tasks | From enrollment to the end of followup after 10 years
  Sound levels include Environmental Sound Levels. Hearing tasks includes Pure Tone Audiometry, Speech in Noise, and Tinnitus matching. This outcome is only among Participants that use Apple Watch.
Change from baseline in abbreviated Pure Tone Audiometry following loud environmental noise notification | From enrollment to the end of followup after 10 years
  This assessment will be for two frequencies (1 kHz and 4 kHz for both ears) tested within 24 hours of acute loud Environmental Sound Level exposure (LEQ equivalent to >97 dBA for >30 minutes). This outcome is only among Participants that use Apple Watch.
Assess reported participant experience | From enrollment to the end of followup after 10 years
  Experience will be assessed via survey delivered with a notification after a prolonged loud environmental sound level exposure (LEQ equivalent to >80 dBA for >40 hours). This outcome is only among Participants that use Apple Watch.
Association between heart rate measures and Headphone Audio Level patterns | From enrollment to the end of followup after 10 years
  This will include heart rate during activity (as assessed by logged Workouts and Active Energy trends by Watch). This outcome is only among participants that use Apple Watch.
Association between heart rate measures and Environmental Sound Level patterns | From enrollment to the end of followup after 10 years
  This includes heart rate during activity (as assessed by logged Workouts and Active Energy trends by Watch). This outcome is only among participants that use Apple Watch.

OTHER OUTCOMES:
Impact of hearing ability on other related aspects of health | From enrollment to the end of followup after 10 years
  Health includes things such as activity, cognition, mental health, mobility, sleep, health conditions, and health outcomes.
Assess novel versions of hearing assessments | From enrollment to the end of followup after 10 years
  These assessments will be delivered using Research app. This may include different variations of speech in noise, pure tone audiometry, and related assessments such as evoked otoacoustic emissions (EOAE).

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Neitzel, PhD, MS, CIH, Principal Investigator — University of Michigan; Lauren M Smith, MS, MPH, Study Director — University of Michigan; Joyce M Daniels, MA, Study Chair — University of Michigan
Locations (1):
- University of Michigan School of Public Health, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
N/A - no plan to share

REFERENCES:
- [Background] Smith LM, Wang L, Mazur K, Carchia M, DePalma G, Azimi R, Mravca S, and Neitzel RL. Impacts of COVID-19-related social distancing measures on personal environmental sound exposures. Environmental Research Letters. Oct 2020. 15.10: 104094. https://iopscience.iop.org/article/10.1088/1748-9326/abb494
- [Background] Neitzel RL, Smith L, Wang L, Green G, Block J, Carchia M, Mazur K, DePalma G, Azimi R, Villanueva B. Toward a better understanding of nonoccupational sound exposures and associated health impacts: Methods of the Apple Hearing Study. J Acoust Soc Am. 2022 Mar;151(3):1476. doi: 10.1121/10.0009620. PMID 35364926
- See also: UM Study Website — https://sph.umich.edu/applehearingstudy/